CLINICAL TRIAL: NCT07031492
Title: Beyond Hybrid Artificial Pancreas Systems: Relieving Carb Counting Via Flexible-userinteraction Multiple-input Control Architectures
Brief Title: Relieving Carb Counting Via Flexible-userinteraction Multiple-input Control Architectures
Acronym: FLEX-AP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLEX-AP
Record Dates: First submitted 2025-05-16; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: T1DM - Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The intented purpose of FLEX-AP is to improve the glycemic control of patients with Type 1 Diabetes (T1D) against events of unannounced meals by automating the calculation of the regulatory action (insulin infusion). To this end, FLEX-AP will periodically ( each 5 min) receive the glucose value fron a continuous glucose monitoring (CGM). Then, FLEX-AP´s control algorithm will use the received glucose value (input to the algorithm) to compute a new value of insulin infusion. Then, it will send the calculated insuline infusion to the pump. Complementarily, it will alert users to hyperglycemia an d hypoglicemia.
  This is a preliminary, exploratory non-randomized, longitudinal, crossover study involving patients with T1D who are habitual userss of the Minimed 780G hybrid closed-loop system. This study consists of two sequentials phases, starting wiht the Minimed 780G hybrid closed-loop system and transitioning to the FLEX-AP system, with no randomization of treatment orde
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation of FLEX-AP system (Experimental): This is a preliminary, exploratory non-randomized, longitudinal, crossover study involving patients with T1D who are habitual userss of the Minimed 780G hybrid closed-loop system. This study consists of two sequentials phases, starting wiht the Minimed 780G hybrid closed-loop system and transitioning to the FLEX-AP system, with no randomization of treatment order.
  Interventions: Device: FLEX-AP system will be implemented to T1D patients

INTERVENTIONS:
Device: FLEX-AP system will be implemented to T1D patients — A FLEX-AP system will be implemented to T1D patients after they have been given a Minimed 780G hybrid closed-loop system

SUMMARY:
Developing algorithms for Automated Insulin Delivery (AID) systems that alleviate the burden of meal announcements, culminating in the FLEX-AP system. This fully automated artificial pancreas system is designed to operate without meal or exercise announcements while allowing for optional user input. FLEX-APaims to achieve a balance between glycemic control and user quality of life by incorporating user preferences into its operation.

The FLEX-AP system features a flexible control architecture tailored to handle unannounced meals and exercise. It also allows for optional meal announcements and offers guidance for mitigating hypoglycemia, such as counterregulatory actions like rescue carbohydrate intake for patients who prefer it. The proposed benefit of FLEX-AP is to improve glycemic control while respecting individual preferences, which sets it apart from existing AID systems.

DETAILED DESCRIPTION:
Although AID systems have significantly advanced, carbohydrate counting remains a burdensome and error-prone task for patients, often leading to suboptimal postprandial glycemic control. Furthermore, even with accurate carbohydrate estimation, other macronutrients impact glycemic responses, complicating management. Hybrid AID systems that rely on meal announcements to manage glycemic excursions, but theses exhibit a limited efficacy when managing moderate-to-large unannounced meals, underscoring the need for systems with improved adaptability and functionality.

The FLEX-AP system features a flexible control architecture tailored to handle unannounced meals and exercise. It also allows for optional meal announcements and offers guidance for mitigating hypoglycemia, such as counterregulatory actions like rescue carbohydrate intake for patients who prefer it. The proposed benefit of FLEX-AP is to improve glycemic control while respecting individual preferences, which sets it apart from existing AID systems.

The first clinical trial that uses the FLEX-AP system (NCT06082973) was approved by the Spanish regulatory agency (AEMPS) in April 2024 and it is currently ongoing. This study evaluates the FLEX-AP in a hospital setting under unannounced exercise challenges to assess the functionality of counter-regulatory actions recommendation, comparing rescue carbohydrates versus mini-doses of glucagon.

The rationale of this study is to advance the evaluation of the FLEX-AP system for fully automated postprandial glucose control under inpatient and outpatient conditions, going beyond in-silico studies. This study is designed to determine safety and efficacy of the FLEX-AP system in a controlled ambulatory condition, emulating real-life conditions. Patients will operate the system as fully-automated for meals under 70 grams of carbohydrates, announcing larger meals as safety measure in this first ambulatory study. This study will provide essential insights for engineers to understand complex meal dynamics better, facilitating further refinement of the FLEX-AP algorithm required for pivotal studies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years inclusive.
* T1D as per the American Diabetes Association classification for >12 months prior to the screening visit.
* Minimed 780G®-hybrid closed-loop system users for at least 6 months. Use of automatic mode (Smartguard) > 80% of the time.
* A1c level below 9.0% at Screening visit.
* Assessment of albuminuria and retinal tests, which should have yielded negative results for advanced medical complications.
* Willing and able to adhere to the study protocol

Exclusion Criteria:

* Not having met the previous criteria for inclusion.
* Females who are pregnant or intend to become pregnant during the study period; a positive pregnancy test at screening will result in exclusion.
* Breastfeeding.
* Use of any non-insulin glucose-lowering therapy within three months prior to study initiation.
* Presence of moderate/severe renal impairment, defined as an estimated glomerular filtration rate (eGFR) <40 mL/min/1.73 m².
* History of severe hypoglycemia (defined as coma or convulsion requiring assistance from others) or diabetic ketoacidosis in the six months prior to study initiation.
* Hypoglycemia unawareness (defined as Clarke Test score greater than 3).
* Occurrence of an acute cardiovascular event (e.g., myocardial infarction, unstable angina, stroke) within twelve months prior to study initiation.
* History of drug or alcohol abuse. History of any active or suspected malignancy.
* Clinically significant microvascular complications (such as macroalbuminuria, preproliferative and proliferative retinopathy), cardiovascular, hepatic, neurological, endocrine, or other systemic conditions, apart from T1D, that may hinder the implementation of the clinical study protocol or the interpretation of study results.
* Diabetic gastroparesis.
* Scheduled surgery during the study period.
* Adherence to a very low carbohydrate diet, defined as a carbohydrate intake of less than 40 grams per day.
* Presence of any comorbid medical or psychological condition deemed by the investigators to render the individual unsuitable for study participation.
* Known allergy to insulin NovoRapid.
* Regular practice of competitive or very high intensity physical activity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the FLEX-AP system | 4 weeks
  Percentage of time spent in target sensor glucose range (70-180 mg/dL, Time in range (TIR)) during the FLEX-AP controlled ambulatory phase in Automatic mode.
Safety of the FLEX-AP system | 4 weeks
  To assess the safety of the FLEX-AP system in a controlled ambulatory setting simulating real-life conditions:Number of symptomatic hypoglycemia events, Number of severe hypoglycemia events, Episodes of diabetic ketoacidosis (DKA) or ketosis, Technical issues related to the insulin pump and dermatological issues related to device use.

SECONDARY OUTCOMES:
Continuous glucose monitoring (CGM) data during the FLEX-AP controlled ambulatory phase in automatic mode will be analyzed according to the following standardized CGM metrics for clinical trials. | 4 weeks
  1) Percentage of participants able to maintain TIR>70% (70-180 mg/dL). This outcome will be calculated for two time periods: 1) daytime (06:00 - 23:59 hours), and 2) nighttime (00:00 - 05:59 hours).
Continuous glucose monitoring (CGM) data during the FLEX-AP controlled ambulatory phase in automatic mode will be analyzed according to the following standardized CGM metrics for clinical trials. | 4 weeks
  2) TIR, defined as % CGM time 70-140 mg/dL. This outcomes will be calculated for two time periods: 1) daytime (06:00 - 23:59 hours), and 2) night time (00:00 - 05:59 hours).
Continuous glucose monitoring (CGM) data during the FLEX-AP controlled ambulatory phase in automatic mode will be analyzed according to the following standardized CGM metrics for clinical trials. | 4 weeks
  3) % CGM time in Level 1 hypoglycemia (CGM <70 mg/dL and > 54 mg/dL). This outcomes will be calculated for two time periods: 1) daytime (06:00 - 23:59 hours), and 2) night time (00:00 - 05:59 hours).
Continuous glucose monitoring (CGM) data during the FLEX-AP controlled ambulatory phase in automatic mode will be analyzed according to the following standardized CGM metrics for clinical trials. | 4 weeks
  4) % CGM time in Level 2 hypoglycemia (CGM ≤ 54 mg/dL). This outcome will be calculated for two time periods: 1) daytime (06:00 - 23:59 hours), and 2) night time (00:00 - 05:59 hours).
Continuous glucose monitoring (CGM) data during the FLEX-AP controlled ambulatory phase in automatic mode will be analyzed according to the following standardized CGM metrics for clinical trials. | 4 weeks
  5) % CGM time in Level 1 hyperglycemia (CGM >180 mg/dL and ≤ 250 mg/dL). This outcome will be calculated for two time periods: 1) daytime (06:00 - 23:59 hours), and 2) night time (00:00 - 05:59 hours).
Continuous glucose monitoring (CGM) data during the FLEX-AP controlled ambulatory phase in automatic mode will be analyzed according to the following standardized CGM metrics for clinical trials. | 4 weeks
  6) % CGM time in Level 2 hyperglycemia (CGM > 250 mg/dL). This outcome will be calculated for two time periods: 1) daytime (06:00 - 23:59 hours), and 2) night time (00:00 - 05:59 hours).
Continuous glucose monitoring (CGM) data during the FLEX-AP controlled ambulatory phase in automatic mode will be analyzed according to the following standardized CGM metrics for clinical trials. | 4 weeks
  7) Mean sensor glucose and glucose variability (expressed primarily as coefficient of variation and second as an SD). This outcome will be calculated for two time periods: 1) daytime (06:00 - 23:59 hours), and 2) night time (00:00 - 05:59 hours).
The glycemic outcome within the postprandial period will be assessed, in an exploratory analysis, with the 5-h postprandial percent TIR (70-180 mg/dL) | 4 weeks
  This will be conducted for the unannounced and announced breakfast in the FLEX-AP controlled hospital phase, comparing with their counterparts in the Minimed 780G® controlled hospital phase. Postprandial periods assessment during the FLEX-AP controlled ambulatory phase in Automatic mode will also be conducted.
The glycemic outcome within the postprandial period will be assessed, in an exploratory analysis, the 5-h postprandial glucose incremental area under the curve. | 4 weeks
  This will be conducted for the unannounced and announced breakfast in the FLEX-AP controlled hospital phase, comparing with their counterparts in the Minimed 780G® controlled hospital phase. Postprandial periods assessment during the FLEX-AP controlled ambulatory phase in Automatic mode will also be conducted.
Efficacy of the FLEX-AP system | 4 weeks
  Total daily insulin during the FLEX-AP controlled ambulatory phase in Automatic mode will be also calculated for exploratory purposes. Active sustance: aspart, formulation: cartridge containing 3ml of insulin solution: 100 IU/ ml, 1 U equals 6 nmol
Efficacy of the FLEX-AP system | 4 weeks
  The number of manual correction boluses during the FLEX-AP controlled ambulatory phase in Automatic mode will be also calculated for exploratory purposes. Modifications of insulin dose according glucose range ( 70-180 mg/dl)
Efficacy of the FLEX-AP system | 4 weeks
  Number of unannounced meals during the FLEX-AP controlled ambulatory phase in Automatic mode.
To evaluate the patients perceptions | 4 weeks
  The patient will complete the PROMs assessment questionnaires at the end of the FLEX-AP controlled ambulatory phase in Automatic mode: Perceptions, Ideas, Reflections and Expectations questionnaire (INSPIRE)
To evaluate the patients perceptions | 4 weeks
  The patient will complete the PROMs assessment questionnaires at the end of the FLEX-AP controlled ambulatory phase in Automatic mode: Hypoglycemia Fear Survey (HFS)
To evaluate the patients perceptions | 4 weeks
  The patient will complete the PROMs assessment questionnaires at the end of the FLEX-AP controlled ambulatory phase in Automatic mode: Diabetes Distress Scale (DDS).
To evaluate the patients perceptions | 4 weeks
  The patient will complete the PROMs assessment questionnaires at the end of the FLEX-AP controlled ambulatory phase in Automatic mode: Diabetes Quality of Life (DQoL).
To evaluate the patients perceptions | 4 weeks
  The patient will complete the PROMs assessment questionnaires at the end of the FLEX-AP controlled ambulatory phase in Automatic mode: System Usability Scale (SUS)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Bondia, PhD, Principal Investigator — Universitat Politecnica Valencia, Spain
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

REFERENCES:
- [Background] Shalit R, Minsky N, Laron-Hirsh M, Cohen O, Kurtz N, Roy A, Grosman B, Benedetti A, Tirosh A. Unannounced Meal Challenges Using an Advanced Hybrid Closed-Loop System. Diabetes Technol Ther. 2023 Sep;25(9):579-588. doi: 10.1089/dia.2023.0139. PMID 37335759
- [Background] Tornese G, Carletti C, Giangreco M, Nistico D, Faleschini E, Barbi E. Carbohydrate Tolerance Threshold for Unannounced Snacks in Children and Adolescents With Type 1 Diabetes Using an Advanced Hybrid Closed-Loop System. Diabetes Care. 2022 Jun 2;45(6):1486-1488. doi: 10.2337/dc21-2643. PMID 35522033